CLINICAL TRIAL: NCT02661893
Title: An Open-Label Drug Interaction Study to Assess the Pharmacokinetics of JNJ-42847922 When Administered Alone and in Combination With Rifampin in Healthy Male and Female Subjects
Brief Title: A Drug Interaction Study in Healthy Participants to Assess the Effect of Rifampin on the Pharmacokinetics of JNJ-42847922
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108077; 42847922EDI1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-01-05; First posted 2016-01-25 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42847922; Rifampin; Pharmacokinetics
MeSH Terms: interventions — seltorexant; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-42847922 and Rifampin (Experimental): A single oral dose of 40 milligram (mg) (=2*20 mg) dose of JNJ-42847922 on Day 1; A single oral dose of 40 mg (=2*20 mg) dose of JNJ-42847922 dosed with one oral dose of rifampin 600 mg (2*300 mg) on Day 5; A single oral dose of 40 mg (=2*20 mg) dose of JNJ-42847922 dosed on Day 12, following once daily dosing of rifampin with an oral dose of rifampin 600 mg (2*300 mg) on Days 5-12.
  Interventions: Drug: JNJ-42847922; Drug: Rifampin

INTERVENTIONS:
Drug: JNJ-42847922 — A single oral dose of 40 milligram (mg) (=2*20 mg) dose of JNJ42847922 on Day 1, Day 5 and Day 12.
Drug: Rifampin — Oral dose of rifampin 600 mg (2*300 mg) on Day 5 and once daily dosing of rifampin with an oral dose of rifampin 600 mg (2*300 mg) on Days 5 to 12.

SUMMARY:
The purpose of this study is to assess the effect of single- and multiple-dose of rifampin on the single-dose pharmacokinetics of JNJ-42847922 after oral administration to healthy male and female participants.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, single-center, multiple-dose study in 14 healthy adults. All participants will receive a single oral dose of 40 milligram (mg) JNJ-42847922 on 3 separate occasions: Day 1 (JNJ-42847922 alone), Day 5 (JNJ-42847922 with a single dose of rifampin), and Day 12 (JNJ-42847922 in combination with steady-state rifampin). A daily dose of 600 mg (2 * 300 mg) rifampin will be administered from Day 5 through Day 12. Following JNJ-42847922 dosing, serial blood samples will be collected over 48 hours for the evaluation of plasma concentrations of JNJ-42847922 and its metabolites. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-child-bearing potential between 18 and 60 years of age, inclusive; body mass index (BMI) between 18 and 30 kilogram (kg)/meter^2, inclusive, and body weight of not less than 50 kg who are nonsmokers (current and for past 60 days)

Exclusion Criteria:

* History of or current clinically significant medical illness
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG)
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of the study drug is scheduled until completion of the study
* Received a known inhibitor of cytochrome P450 (CYP) 3A4 or CYP2C9 activity within 28 days or a period less than 5 times the drugs half-life; whichever is longer, before the first dose of the study drug is scheduled

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by maximum plasma concentration (Cmax) on Day 1 | Day 1
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by maximum plasma concentration (Cmax) on Day 5 | Day 5
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by maximum plasma concentration (Cmax) on Day 12 | Day 12
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by Area Under the Plasma Concentration-Time Curve (AUC) on Day 1 | Day 1
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by Area Under the Plasma Concentration-Time Curve (AUC) on Day 5 | Day 5
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.
Pharmacokinetics of JNJ-42847922 and metabolites M12 and M16 as assessed by Area Under the Plasma Concentration-Time Curve (AUC) on Day 12 | Day 12
  Blood samples will be collected after dosing of JNJ-42847922 on each occasion to assess the pharmacokinetics of JNJ-42847922 and metabolites M12, M16 with and without rifampin.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to Day 44
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States